CLINICAL TRIAL: NCT06990308
Title: A Single-center, Patient- and Assessor-blinded, Randomized Controlled Trial to Compare Patient Outcomes Between Deflated and Inflated Cuff Endotracheal Extubations During Scheduled, Non-airway Surgery in Healthy Adults
Brief Title: Deflated and Inflated Cuff Endotracheal Extubations
Acronym: DICEE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Naval Medical Center Camp Lejeune (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Lee, Staff Anesthesiologist, Naval Medical Center Camp Lejeune
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCCL.2025.0007
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia Airway Management; Respiratory Complications
Keywords: General Endotracheal Anesthesia; Deflated Cuff Extubation; Inflated Cuff Extubation; Microaspiration; Airway Contamination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inflated Cuff Arm: 44 (Experimental): Extubation with an inflated endotracheal tube cuff
  Interventions: Procedure: Inflated Cuff Extubation
- Deflated Cuff Arm: 44 (Active Comparator): Extubation with a deflated endotracheal tube cuff
  Interventions: Procedure: Deflated Cuff Extubation

INTERVENTIONS:
Procedure: Inflated Cuff Extubation — The adjustable pressure limiting valve will be set to 20 centimeters water pressure. To blind the Anesthesiologist Associate Investigator from the patient's group allocation, sham deflation of the endotracheal tube cuff pilot balloon will be performed with a 10 milliliter syringe. The endotracheal tube will be withdrawn into an opaque blue towel while the reservoir bag is simultaneously compressed to generate at least 20 centimeters water pressure positive airway pressure. In the rare event significant resistance is met with attempted extubation, the principal investigator will deflate the cuff in one milliliter increments until extubation is possible. This process does not unblind the Anesthesiologist Associate Investigator.
  Arms: Inflated Cuff Arm: 44
Procedure: Deflated Cuff Extubation — The adjustable pressure-limiting valve will be set to 20 centimeters water pressure. All air will be removed from the endotracheal tube cuff pilot balloon with a 10 milliliter syringe. The endotracheal tube will be withdrawn into an opaque blue towel, to prevent the Anesthesiologist Associate Investigator from identifying the patient's allocation, while the reservoir bag is simultaneously compressed to generate at least 20 centimeters water pressure positive airway pressure.
  Arms: Deflated Cuff Arm: 44

SUMMARY:
General anesthesia is a treatment with medicine to make a patient unconscious for surgery. This is sometimes called "being put to sleep" or "being put under." Most of the time, a breathing tube is used to help a machine breathe for patients. The breathing tube has a cuff, which is like a small balloon. After the breathing tube is placed, the cuff is inflated. This keeps the breathing tube in place and keeps fluids like saliva and stomach juices from getting into the windpipe and lungs. When a breathing tube is removed, that is called extubation.

Normally, doctors deflate the cuff before removing the breathing tube. This is called deflated cuff extubation. Some doctors worry that keeping the cuff inflated while it is removed can damage the throat or vocal cords. However, some doctors keep the cuff inflated when removing the breathing tube. This is called inflated cuff extubation. These doctors think that keeping the cuff inflated can help keep fluids from entering the airway.

Doctors have not studied if deflated cuff extubation is better or worse than inflated cuff extubation. The goal of this study is to see which type of extubation is better at keeping fluids from getting in the airway.

Participants who are part of this study will get general anesthesia and have surgery as planned. Near the end of surgery, a small amount of liquid is placed at the back of a participant's mouth. This liquid is called contrast material, and it is like a dye. The contrast material will help determine if any liquid enters the windpipe or lungs. Then, contrast material is removed, along with any other fluids, using normal methods.

When it is safe to take the breathing tube out, a deflated cuff extubation or an inflated cuff extubation will be performed. This decision will be made at random, like by the flip of a coin. Information will be collected about participants, the surgery, and how well a participant is breathing. After surgery, a chest x-ray will be taken to see if any of the contrast material is in the windpipe or lungs. Otherwise, everything else after surgery would be normal. 24 to 48 hours after surgery, a member of the research team will ask about any symptoms a participant may have, like sore throat or a hoarse voice. Research would conclude at that time.

DETAILED DESCRIPTION:
The current standard anesthetic practice for extubation is to deflate the endotracheal tube cuff using a syringe prior to extubation. While commonplace and nearly universally accepted, this practice is not based on evidence from randomized controlled trials but is instead due to concern for laryngeal or vocal cord injury and arytenoid cartilage dislocation. However, no publications exist in the medical literature that attribute laryngeal trauma directly to inflated cuff endotracheal tube extubation, as opposed to the process of extubation in general. To the contrary, case reports that describe peri operative extubation with unintentionally inflated cuffs all note the absence of negative outcome.

Alternatively, extubation with an inflated endotracheal tube cuff has been advocated as a technique to reduce airway complications in human and veterinary medicine. Tracheal aspiration, even micro-aspiration by oropharyngeal secretions, may increase the risk of pneumonia and other pulmonary complications. Based on an animal model, inflated cuff extubation may reduce airway contamination by oropharyngeal fluid. Additionally, leaving the endotracheal tube cuff inflated may effectively generate a vital capacity breath during extubation, maximizing oxygen reserves and facilitating a secretion-clearing cough. These theorized advantages may prolong the time to which supplemental oxygen is required as well as decrease airway/respiratory complications in the immediate post-extubation period. Within the intensive care setting, unplanned extubation (including accidental extubation and self-extubation) occurs at a rate of 3% to 16% of intubated patients or 0.1 to 3.6 per 100 days of mechanical ventilation. Estimates of national hospitalizations requiring mechanical ventilation approach 800,000, thereby placing the estimated number of unplanned extubations between 24,000 and 128,000. Presumably, the majority of these unplanned extubations are with inflated cuffs, and yet still no epidemic of laryngeal trauma from inflated cuff extubation exists. Furthermore, there have been no significant differences in laryngeal complications reported between planned and unplanned extubation in the intensive care population, suggesting that it is the endotracheal tube itself (and the process of placing it) that confers the risk of laryngeal complications, rather than the circumstances of its removal.

Though several providers have published their success with inflated cuff extubation, to date no prospective, randomized controlled trial has been performed directly comparing these two techniques. This study proposes to evaluate the effect of inflated cuff extubation on airway contamination by oropharyngeal material, extubation quality, post-extubation oxygenation, and laryngeal symptoms compared to the standard technique of deflated cuff extubation.

To assess the difference in aspiration rates between deflated and inflated cuff extubation, radio-opaque contrast material will be introduced into the oropharynx of intubated patients while under general anesthesia. The presence of this radio-opaque contrast at or below the level of the carina will be assessed with a chest radiograph taken postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 50 years old
* Scheduled for surgery, not of the airway, head, or neck, with anticipated case duration of less than 3 hours
* American Society of Anesthesiologists (ASA) Physical Status Classification of 1 to 3

Exclusion Criteria:

* Emergent surgery, or surgery requiring prone, sitting or lateral positioning
* Pre-existing laryngeal pathology, obstructive pulmonary disease, pulmonary hypertension, interstitial lung disease, active respiratory infection, recent pneumonia, uncontrolled asthma, or uncontrolled gastroesophageal reflux disease
* Known difficulties with general anesthesia, such as prior anaphylactic reaction, difficult intubation or mask ventilation
* Known allergy to iohexol or a previous severe reaction to any contrast agents
* Unfavorable airway examination, such as Mallampati 4, limited mouth opening, and/or inability to extend neck
* Non-compliance with ASA Practice Guidelines for Preoperative Fasting
* Pregnancy
* Enrollment in another anesthesiology or surgery related interventional research study
* Surgeries scheduled on Friday or a day immediately prior to a holiday

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Airway Contamination | 0-30 minutes after arrival in the Post Anesthesia Care Unit
  Number of patients with presence of radio-opaque contrast material at or below the level of the carina on portable chest radiograph (yes/no)

SECONDARY OUTCOMES:
Hypoxemia | 0 to 6 minutes after tracheal extubation
  Yes/No as defined by Arterial Saturation Pulse Oximeter (SpO2) reading of <95%
  None Spo2 ≥ 95% Mild Spo2 91% - 94% Moderate Spo2 86% - 90% Severe Spo2 80% - 85% Critical Spo2 ≤ 79%
  Lowest SpO2 reading will be recorded
Need for Supplemental Oxygen | 0-6 minutes after tracheal extubation
  Arterial Desaturation to <95% SpO2 requiring oxygen supplementation Yes/No Time (in seconds)
Cough | 0 to 6 minutes after tracheal extubation
  5-point Modified Minogue Scale (0-4)
Obstruction | 0 to 6 minutes after tracheal extubation
  Yes/No
Stridor | 0 to 6 minutes after tracheal extubation
  Yes/No
Bronchospasm | 0 to 6 minutes after tracheal extubation
  Yes/No
Laryngospasm | 0 to 6 minutes after tracheal extubation
  Yes/No
Aspiration | 0 to 6 minutes after tracheal extubation
  Yes/No
Sore Throat | 24-48 hours postoperatively
  4-point Likert Scale, 0-3
Cough | 24-48 hours postoperatively
  4-point Simplified Cough Score, 0-3
Voice Quality | 24-48 hours postoperatively
  GRBAS scale: Grade (0-3), Roughness (0-3), Breathiness (0-3), Aesthenia (0-3), Strain (0-3)
Dysphagia | 24-48 hours postoperatively
  4-point Bazaz Dysphagia Score (0-3)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Lee, MD, Principal Investigator — Naval Medical Center Camp Lejeune
Locations (1):
- Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participant data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol, SAP, ICF will be available beginning 24APR2025 indefinitely, de-identified individual participant data will be available approximately SEP2026-SEP2033
Access Criteria: Medical and research professionals by request

REFERENCES:
- [Background] Lin EC. Radiation risk from medical imaging. Mayo Clin Proc. 2010 Dec;85(12):1142-6; quiz 1146. doi: 10.4065/mcp.2010.0260. PMID 21123642
- [Background] Lasser EC, Lyon SG, Berry CC. Reports on contrast media reactions: analysis of data from reports to the U.S. Food and Drug Administration. Radiology. 1997 Jun;203(3):605-10. doi: 10.1148/radiology.203.3.9169676.
- [Background] Caro JJ, Trindade E, McGregor M. The risks of death and of severe nonfatal reactions with high- vs low-osmolality contrast media: a meta-analysis. AJR Am J Roentgenol. 1991 Apr;156(4):825-32. doi: 10.2214/ajr.156.4.1825900.
- [Background] Wolf GL, Arenson RL, Cross AP. A prospective trial of ionic vs nonionic contrast agents in routine clinical practice: comparison of adverse effects. AJR Am J Roentgenol. 1989 May;152(5):939-44. doi: 10.2214/ajr.152.5.939. PMID 2495706
- [Background] Katayama H, Yamaguchi K, Kozuka T, Takashima T, Seez P, Matsuura K. Adverse reactions to ionic and nonionic contrast media. A report from the Japanese Committee on the Safety of Contrast Media. Radiology. 1990 Jun;175(3):621-8. doi: 10.1148/radiology.175.3.2343107.
- [Background] Molfenter SM, Amin MR, Balou M, Herzberg EG, Frempong-Boadu A. A scoping review of the methods used to capture dysphagia after anterior cervical discectomy and fusion: the need for a paradigm shift. Eur Spine J. 2023 Mar;32(3):969-976. doi: 10.1007/s00586-022-07515-1. Epub 2023 Jan 10. PMID 36625955
- [Background] De Bodt MS, Wuyts FL, Van de Heyning PH, Croux C. Test-retest study of the GRBAS scale: influence of experience and professional background on perceptual rating of voice quality. J Voice. 1997 Mar;11(1):74-80. doi: 10.1016/s0892-1997(97)80026-4. PMID 9075179
- [Background] Ghio A, Revis J, Smithson-Barriere D, Jarze S, Giovanni A. Reliability and Correlations Between Overall Severity, Roughness and Breathiness in the Perception of Dysphonic Voices: Investigating Cognitive Aspects. J Voice. 2024 Jan;38(1):136-143. doi: 10.1016/j.jvoice.2021.07.010. Epub 2021 Aug 25. PMID 34452778
- [Background] Tung A, Fergusson NA, Ng N, Hu V, Dormuth C, Griesdale DGE. Pharmacological methods for reducing coughing on emergence from elective surgery after general anesthesia with endotracheal intubation: protocol for a systematic review of common medications and network meta-analysis. Syst Rev. 2019 Jan 24;8(1):32. doi: 10.1186/s13643-019-0947-2. PMID 30678727
- [Background] Minogue SC, Ralph J, Lampa MJ. Laryngotracheal topicalization with lidocaine before intubation decreases the incidence of coughing on emergence from general anesthesia. Anesth Analg. 2004 Oct;99(4):1253-1257. doi: 10.1213/01.ANE.0000132779.27085.52. PMID 15385385
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Dejonckere PH, Wieneke GH. GRBAS-scaling of pathological voices: reliability, clinical relevance and differentiated correlation with acoustic measurements, especially with central measurements. Proceedings of the 22nd IALP Congress. Hannover, Germany: 1992.
- [Background] Hirano M. Clinical examination of voice. New York: Springer Verlag, 1981:81-4.
- [Background] Lin R, Zhu L, Pan X. Validation of the simplified cough symptom score in non-small cell lung cancer patients after surgery. Gen Thorac Cardiovasc Surg. 2022 Aug;70(8):735-739. doi: 10.1007/s11748-022-01791-w. Epub 2022 Feb 28. PMID 35224703
- [Background] Lai K. Chinese National Guidelines on Diagnosis and Management of Cough: consensus and controversy. J Thorac Dis. 2014 Oct;6(Suppl 7):S683-8. doi: 10.3978/j.issn.2072-1439.2014.10.06. No abstract available. PMID 25383201
- [Background] Sivanandam LK, Verghese RJ, Balan S, Balamurugesan K. Accidental iohexol bronchography. BMJ Case Rep. 2021 Aug 5;14(8):e244942. doi: 10.1136/bcr-2021-244942. No abstract available. PMID 34353841
- [Background] Sarkar P, Patel N, Chusid J, Shah R, Talwar A. The role of computed tomography bronchography in the management of bronchopleural fistulas. J Thorac Imaging. 2010 Feb;25(1):W10-3. doi: 10.1097/RTI.0b013e31819d12f1. PMID 20160584
- [Background] MacIntyre P, Peacock C, Gordon I, Mok Q. Use of tracheobronchography as a diagnostic tool in ventilator-dependent infants. Crit Care Med. 1998 Apr;26(4):755-9. doi: 10.1097/00003246-199804000-00028. PMID 9559615
- [Background] Little AF, Phelan EM, Boldt DW, Brown TC. Paediatric tracheobronchomalacia and its assessment by tracheobronchography. Australas Radiol. 1996 Nov;40(4):398-403. doi: 10.1111/j.1440-1673.1996.tb00434.x. PMID 8996899
- [Background] Deutsch ES, Smergel E, Crisci K, Panitch H. Tracheobronchography in children. Laryngoscope. 1996 Oct;106(10):1248-54. doi: 10.1097/00005537-199610000-00016. PMID 8849796
- [Background] Hwang CH. Swallowing study using water-soluble contrast agents may increase aspiration sensitivity and antedate oral feeding without respiratory and drug complications: A STROBE-compliant prospective, observational, case-control trial. Medicine (Baltimore). 2022 Jul 8;101(27):e29422. doi: 10.1097/MD.0000000000029422. PMID 35801762
- [Background] Harris JA, Bartelt D, Campion M, Gayler BW, Jones B, Hayes A, Haynos J, Herbick S, Kling T, Lingaraj A, Singer M, Starmer H, Smith C, Webster K. The use of low-osmolar water-soluble contrast in videofluoroscopic swallowing exams. Dysphagia. 2013 Dec;28(4):520-7. doi: 10.1007/s00455-013-9462-0. Epub 2013 Mar 26. PMID 23529533
- [Background] Sun J, Li Z. Study on the Correlation between Barium Radiography and Pulmonary Infection rate in the Evaluation of Swallowing Function. Clinics (Sao Paulo). 2018;73:e182. doi: 10.6061/clinics/2018/e182. Epub 2018 Jun 18. PMID 29924183
- [Background] Morcos SK. Review article: Effects of radiographic contrast media on the lung. Br J Radiol. 2003 May;76(905):290-5. doi: 10.1259/bjr/54892465. PMID 12763943
- [Background] Claussen D. Omnipaque (iohexol). Gastroenterol Nurs. 1992 Jun;14(6):307-9. doi: 10.1097/00001610-199206000-00007. PMID 1623033
- [Background] Brick SH, Caroline DF, Lev-Toaff AS, Friedman AC, Grumbach K, Radecki PD. Esophageal disruption: evaluation with iohexol esophagography. Radiology. 1988 Oct;169(1):141-3. doi: 10.1148/radiology.169.1.3420250.
- [Background] Yan GW, Deng JF, Bhetuwal A, Yang GQ, Fu QS, Chen H, Hu N, Zeng H, Fan XP, Yan GW, Wu XL. A case report and literature review of barium sulphate aspiration during upper gastrointestinal examination. Medicine (Baltimore). 2017 Nov;96(47):e8821. doi: 10.1097/MD.0000000000008821. PMID 29381987
- [Background] Cork RC, Depa RM, Standen JR. Prospective comparison of use of the laryngeal mask and endotracheal tube for ambulatory surgery. Anesth Analg. 1994 Oct;79(4):719-27. doi: 10.1213/00000539-199410000-00018. PMID 7943782
- [Background] Mraovic B, Hipszer B, Loeum C, Andonakakis A, Joseph J. Evaluation of continuous aspiration of subglottic secretions in prevention of microaspiration during general anesthesia: a randomized controlled pilot study. Croat Med J. 2022 Dec 31;63(6):553-563. doi: 10.3325/cmj.2022.63.553. PMID 36597567
- [Background] Mehta S. The risk of aspiration in presence of cuffed endotracheal tubes. Br J Anaesth. 1972 Jun;44(6):601-5. doi: 10.1093/bja/44.6.601. No abstract available. PMID 5045553
- [Background] Whiffler K, Andrew WK, Thomas RG. The hazardous cuffed endotracheal tube--aspiration and extubation. S Afr Med J. 1982 Feb 13;61(7):240-1. PMID 7058448
- [Result] Atkins PM, Mion LC, Mendelson W, Palmer RM, Slomka J, Franko T. Characteristics and outcomes of patients who self-extubate from ventilatory support: a case-control study. Chest. 1997 Nov 5;112(5):1317-23. doi: 10.1378/chest.112.5.1317. PMID 9367475
- [Result] Boulain T. Unplanned extubations in the adult intensive care unit: a prospective multicenter study. Association des Reanimateurs du Centre-Ouest. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1131-7. doi: 10.1164/ajrccm.157.4.9702083. PMID 9563730
- [Result] Wunsch H, Linde-Zwirble WT, Angus DC, Hartman ME, Milbrandt EB, Kahn JM. The epidemiology of mechanical ventilation use in the United States. Crit Care Med. 2010 Oct;38(10):1947-53. doi: 10.1097/CCM.0b013e3181ef4460. PMID 20639743
- [Result] da Silva PS, Fonseca MC. Unplanned endotracheal extubations in the intensive care unit: systematic review, critical appraisal, and evidence-based recommendations. Anesth Analg. 2012 May;114(5):1003-14. doi: 10.1213/ANE.0b013e31824b0296. Epub 2012 Feb 24. PMID 22366845
- [Result] Kiekkas P, Aretha D, Panteli E, Baltopoulos GI, Filos KS. Unplanned extubation in critically ill adults: clinical review. Nurs Crit Care. 2013 May;18(3):123-34. doi: 10.1111/j.1478-5153.2012.00542.x. Epub 2012 Nov 22. PMID 23577947
- [Result] de Groot RI, Dekkers OM, Herold IH, de Jonge E, Arbous MS. Risk factors and outcomes after unplanned extubations on the ICU: a case-control study. Crit Care. 2011;15(1):R19. doi: 10.1186/cc9964. Epub 2011 Jan 13. PMID 21232123
- [Result] Cosentino C, Fama M, Foa C, Bromuri G, Giannini S, Saraceno M, Spagnoletta A, Tenkue M, Trevisi E, Sarli L. Unplanned Extubations in Intensive Care Unit: evidences for risk factors. A literature review. Acta Biomed. 2017 Nov 30;88(5S):55-65. doi: 10.23750/abm.v88i5-S.6869. PMID 29189706
- [Result] Baftiu N, Krasniqi I, Haxhirexha K, Domi R. Survey about the Extubation Practice among Anaesthesiologists in Kosovo. Open Access Maced J Med Sci. 2018 Feb 12;6(2):350-354. doi: 10.3889/oamjms.2018.083. eCollection 2018 Feb 15. PMID 29531602
- [Result] Vance A, Hofmeister EH, Laas C, Williams J. The effects of extubation with an inflated versus deflated endotracheal tube cuff on endotracheal fluid volume in the dog. Vet Anaesth Analg. 2011 May;38(3):203-7. doi: 10.1111/j.1467-2995.2011.00610.x. PMID 21492385
- [Result] Ephgrave KS, Kleiman-Wexler R, Pfaller M, Booth B, Werkmeister L, Young S. Postoperative pneumonia: a prospective study of risk factors and morbidity. Surgery. 1993 Oct;114(4):815-9; discussion 819-21. PMID 8211699
- [Result] Brown C. Endotracheal intubation in the dog. Lab Anim (NY). 2007 Feb;36(2):23-4. doi: 10.1038/laban0207-23. PMID 17245385
- [Result] Priebe HJ. Could "safe practice" be compromising safe practice? Should anesthetists have to deflate the cuff of the endotracheal tube before extubation? Minerva Anestesiol. 2016 Feb;82(2):236-9. Epub 2015 Jul 1. PMID 26126979
- [Result] Shamsai J. A new technique for removal of endotracheal tube. Anesth Analg. 2006 Oct;103(4):1040. doi: 10.1213/01.ane.0000239021.80428.cb. No abstract available. PMID 17000831
- [Result] Hulme J, Agarwal S. Failure to deflate an endotracheal cuff. Acta Anaesthesiol Scand. 2008 May;52(5):719. doi: 10.1111/j.1399-6576.2007.01467.x. No abstract available. PMID 18419730
- [Result] Sriramka B, Natarajan A, Sharma K, Zubair S. Failed endotracheal tube cuff deflation due to unusual kinking of inflation tube. J Dent Anesth Pain Med. 2023 Aug;23(4):241-243. doi: 10.17245/jdapm.2023.23.4.241. Epub 2023 Jul 29. No abstract available. PMID 37559664
- [Result] Kamata M, Hakim M, Tobias JD. Residual volume in the cuff of the endotracheal tube when the pilot balloon is torn off instead of deflated using a syringe. Int J Pediatr Otorhinolaryngol. 2016 Jul;86:15-8. doi: 10.1016/j.ijporl.2016.04.012. Epub 2016 Apr 12. PMID 27260572
- [Result] Suman S, Ganjoo P, Tandon MS. Difficult extubation due to failure of an endotracheal tube cuff deflation. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):141-2. No abstract available. PMID 21804739
- [Result] Saidman LJ. Where is the evidence? Anesth Analg. 2007 Jul;105(1):285. doi: 10.1213/01.ane.0000278606.10006.fa. No abstract available. PMID 17578998
- [Result] Cooper RM, O'Sullivan E, Popat M, Behringer E, Hagberg CA. Difficult Airway Society guidelines for the management of tracheal extubation. Anaesthesia. 2013 Feb;68(2):217. doi: 10.1111/anae.12139. No abstract available. PMID 23298360

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT06990308/Prot_SAP_ICF_000.pdf